CLINICAL TRIAL: NCT01937325
Title: Airway Infection, Inflammatory Markers and Exercise Capacity in Patients With Cystic Fibrosis and at Least One G551D Mutation Taking VX770 (Ivacaftor)
Brief Title: CPET in CF Patients With One G551D Mutation Taking VX770
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, John Wilson, Head CF Service, The Alfred
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CPET in CF
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Cystic Fibrosis
Keywords: Eligible CF patients with G551D gene mutation
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ivacaftor (Active Comparator): 150mg orally twice daily
  Interventions: Drug: ivacaftor
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ivacaftor — active arm
  Other Names: Kalydeco
  Arms: Ivacaftor
Drug: placebo — active arm
  Other Names: ivacaftor matched placebo
  Arms: Placebo

SUMMARY:
Ivacaftor will restore CFTR function in treated CF patients with the G551D mutation. Improvement in ventilation, salt balance and well-being will contribute to better exercise capacity at all levels of lung function. While potential improvements may be variable across the spectrum of lung function, even small gains at low levels of FEV1 may have significant benefit for some subjects.

DETAILED DESCRIPTION:
The Alfred CF Service is ready to initiate therapy with VX-770 in it's cohort. Investigators therefore have an opportunity to examine correlates between improvements in lung function, exercise capacity, inflammatory markers and indices of wellbeing in CF that may not be repeatable in a single cohort.

Investigators propose a double-blind, placebo-controlled cross-over study of 20 patients currently awaiting initiation of ivacaftor therapy. Patients enrolled in the study will be asked to undergo screening (day -28), and baseline assessments (day 0) and re-assessment studies (day 28) after treatment period 1, followed by baseline assessment at the beginning of treatment period 2 (day 56) and at the conclusion of treatment period 2 (day 84). A further assessment (day 224) will be performed 140 (+/-7) days following commencement on open label Ivacaftor.

After satisfying eligibility criteria, subjects will be randomly assigned to initial active treatment or placebo following a 4 week run-in period. After completion of period 1 and a 4 week washout period, subjects will cross-over to the alternative treatment. After 4 weeks of period 2, subjects will undergo final assessment as shown in the diagram below. However participants choosing not to continue taking ivacaftor in a Named Patient Program or another similar program run by Vertex Pharmaceuticals, Inc., ('Vertex'), at the end of the study period will be required to undergo a Safety Follow-Up visit 28 days after the final dose of study drug. Safety Follow-Up assessments will not include the CPET.

ELIGIBILITY:
Inclusion Criteria:

* All participants will have CF proven based on established criteria (sweat test, genotype and phenotype).
* All participants will have at least one copy of the G551D mutation.
* All will be able to perform an exercise study and complete study questionnaires and assessments.
* Age range will be between 16 and 75 years of age.
* Lung function inclusion will be above 25% predicted FEV1.

Exclusion Criteria:

* Participants will not be included if they are unable to complete study assessments or have had a known adverse reaction to Ivacaftor.
* Female participants will be excluded if found to return a positive pregnancy test at screening.
* Participants will be excluded if using St. John's Wort or rifampicin (strong CYP3A inducers).
* Participants with significant liver dysfunction will be excluded (ALT or ALT above 5 times upper limit of normal).

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
exercise capacity | one month, 3 months
  Respiratory exercise testing, including spirometry and V02 max.

SECONDARY OUTCOMES:
Inflammatory profile | One month, 3 months
  Cytokine levels (IL-1β, IL-6, TNFα, IL-8, VEGF & Activin A) determined using cytometric bead analysis and / or ELISA

CONTACTS AND LOCATIONS:
Overall Officials: John Wilson, Principal Investigator — Alfred Health and Monash University
Locations (1):
- The Alfred, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edgeworth D, Keating D, Ellis M, Button B, Williams E, Clark D, Tierney A, Heritier S, Kotsimbos T, Wilson J. Improvement in exercise duration, lung function and well-being in G551D-cystic fibrosis patients: a double-blind, placebo-controlled, randomized, cross-over study with ivacaftor treatment. Clin Sci (Lond). 2017 Jul 16;131(15):2037-2045. doi: 10.1042/CS20170995. Print 2017 Aug 1. PMID 28611235